CLINICAL TRIAL: NCT04581928
Title: Patients Reactions Towards Their Diagnosis as Having COVID-19: A Cohort Study
Brief Title: Patients Reactions Towards Their Diagnosis as Having COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ClinAmygate (Other)
Responsible Party: Principal Investigator, Emad R Issak, Doctor, ClinAmygate
Other Study IDs: PR0020
Record Dates: First submitted 2020-10-06; First posted 2020-10-09 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Highly educated people Low educated people

SUMMARY:
Patients reactions towards their diagnosis as having COVID-19. The effect of patients' reaction toward their prospect management. How this can make many hazards. Also, obstacle and barrier to better management.

DETAILED DESCRIPTION:
Patients reactions towards their diagnosis as having COVID-19. The effect of patients' reaction toward their prospect management. How this can make many hazards. Also, obstacle and barrier to better management.

Different factors affecting the response of people toward their diagnosis as COVID-19

ELIGIBILITY:
Inclusion Criteria:

* COVID-19
* Age 18 years of less

Exclusion Criteria:

* Mental diseases making the communication with them difficult

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All COVID-19 cases
Sampling Method: Non-Probability Sample
Enrollment: 3812 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to recovery | Four weeks
  Time needed to recovery from symptoms of covid-19

CONTACTS AND LOCATIONS:
Overall Officials: Emad R Issak, MD, Principal Investigator — Assalam Clinics
Locations (1):
- Asalam, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual data will not shared as per local regulations

REFERENCES:
- [Result] Wiseman EJ. Denial in the medical interview. JAMA. 1995 Jun 14;273(22):1735; author reply 1735-6. doi: 10.1001/jama.273.22.1735. No abstract available. PMID 7769754